CLINICAL TRIAL: NCT02978001
Title: Insulin Sensitivity, Glucose - and Fat Metabolism in Patients With Psoriasis
Status: Completed | Type: Observational
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Filip Krag Knop, Professor, University Hospital, Gentofte, Copenhagen
Other Study IDs: MetPso
Record Dates: First submitted 2016-11-26; First posted 2016-11-30 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Insulin Sensitivity; Metabolism Disorder
MeSH Terms: conditions — Insulin Resistance; Metabolic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Muscle and fat biopsies. Blood samples.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Patients with Psoriasis: Patients with moderate to severe psoriasis (PASI>8)
  Interventions: Other: Stabile Isotope tracers
- Healthy Control Subjects: Healthy subjects matching the patients with psoriasis regarding age, gender and BMI
  Interventions: Other: Stabile Isotope tracers

INTERVENTIONS:
Other: Stabile Isotope tracers — Non-radioactive tracers used in hyperinsulinaemic euglycaemic clamp
  Other Names: [6,6-D2]glucose, [1,1,2,3,3,-D5]glycerol

SUMMARY:
The pathophysiological mechanisms explaining the association between psoriasis and type 2 diabetes are largely unknown but it has been hypothesized that systemic inflammation found in both psoriasis and type 2 diabetes might play a role. In a recent study hyperinsulinaemic euglycaemic clamps were performed and it showed that normal glucose-tolerant patients with moderate to severe psoriasis had lower whole-body insulin sensitivity during insulin stimulation compared to healthy matched controls. Thus, the increased risk of type 2 diabetes in patients with psoriasis appears to include defects in the glucose metabolism linked to psoriasis itself. However, the methods applied did not allow a detailed characterization of the metabolism in patients with psoriasis. Tracer technique combined with indirect calorimetry has never been applied to study hepatic and whole body insulin sensitivity, and glucose and fat oxidation, during basal conditions or during insulin stimulation in patients with psoriasis.

Aim of study:

The aim of this study is to investigate hepatic and whole body insulin sensitivity and glucose and fat oxidation during both basal and insulin-stimulated conditions in patients with psoriasis.

DETAILED DESCRIPTION:
Background Psoriasis is a chronic immune-mediated inflammatory disease characterized by uncontrolled proliferation of keratinocytes, activated dendritic cells, release of pro-inflammatory cytokines and recruitment of T-cells to the skin. The prevalence of psoriasis is 2-3% worldwide, with similar frequencies in men and women. Psoriasis has been associated with components of the metabolic syndrome, in particular obesity and type 2 diabetes, and patients with psoriasis are at increased risk of developing type 2 diabetes. Obesity is twice as prevalent in patients with psoriasis and patients are at increased risk of developing cardiovascular disease compared to the general population. These co-morbidities are important to recognize or preferably prevent and treat as they might lead to increased mortality.

Type 2 diabetes is a complex metabolic disorder that develops as a consequence of genetic and environmental factors such as inadequate physical activity and obesity. The incidence of type 2 diabetes is increasing worldwide and there is a general agreement that it is caused mainly by the adoption to westernized, sedentary lifestyle. Patients with type 2 diabetes are characterized by decreased peripheral and hepatic insulin sensitivity, beta cell dysfunction and impaired glucose and fat oxidation. Muscle insulin resistance has been proposed to account for as much as 85-90% of the impairment of the peripheral insulin sensitivity (expressed as the total body glucose disposal) in patients with type 2 diabetes during insulin stimulation. Multiple intramyocellular defects have been demonstrated, including impaired glucose transport and phosphorylation, reduced glycogen synthesis, and decreased glucose oxidation as well as proximal defects in the insulin signal transduction system. Similar to psoriasis, systemic inflammation occurs in patients with type 2 diabetes.

The pathophysiological mechanisms explaining the association between psoriasis and type 2 diabetes are largely unknown but it has been hypothesized that systemic inflammation found in both psoriasis and type 2 diabetes might play a role. In a recent study hyperinsulinaemic euglycaemic clamps were made and it showed that normal glucose-tolerant patients with moderate to severe psoriasis had lower whole-body insulin sensitivity during insulin stimulation compared to healthy matched controls. Thus, the increased risk of type 2 diabetes in patients with psoriasis appears to include defects in the glucose metabolism linked to psoriasis itself. However, the methods applied did not allow a detailed characterization of the metabolism in patients with psoriasis. Tracer technique combined with indirect calorimetry has never been applied to study hepatic and whole body insulin sensitivity, and glucose and fat oxidation, during basal conditions or during insulin stimulation in patients with psoriasis.

Methods:

Prior to experimental day 1 and 2 the participants will meet in the morning following a 10 hour fast (including liquids, medication, and tobacco). No alcohol consumption or vigorous physical activities will be permitted 48 hours before the examination, and all participants will be requested to eat carbohydrate-rich diet the previous two days. All experiments will be carried out in the Center for Diabetes Research, Gentofte Hospital, University of Copenhagen, Hellerup, Denmark where the necessary equipment is available.

Experimental day 1: An intravenous glucose tolerance test (IVGTT), and a fibro scan of the liver will be performed and the second experimental day will be scheduled. Time spent during experimental day 1 is approximately 4 hours.

Intravenous glucose tolerance test (IVGTT) will be performed to determine beta cell function. A glucose bolus of 0.3 g/kg body weight will be infused over 1 min at t=0 min. Plasma samples for glucose, C-peptide, insulin and glucagon will be collected at t = -10, - 5, 0, 2, 4, 6, 8, 10, 15, 20 and 30 min.

Body composition is determined prior to Day 2 by DXA scan (Lunar Prodigy Advance GE Healthcare).

Fibro scan will be performed using a Fibroscan 501® (EchoSensTM, Paris, France) to asses fibrosis status and steatosis grade of the liver (23). Hepatic elasticity and thus fibrosis status (expressed as kPa) will be assessed by measuring the transmission speed of the ultrasound based on the principle that the transmission speed of vibrations passing through liver tissue increases when hepatic fibrosis is present. Hepatic steatosis will be assessed by a controlled attenuation parameter (CAP) (expressed as decibel per meter (dB/m)) based on the fact that fat affects ultrasound propagation. A success rate of ≥60% and a ratio of the interquartile range of liver stiffness to the median ≤30% will be considered reliable and used for the final analysis.

Experimental day 2: Hyperinsulinaemic euglycaemic clamp (HEC) combined with stable isotope infusion, muscle and fat biopsies and indirect calorimetry. Time spent during experimental day 1 is approximately 7 hours.

Following emptying of the urine bladder, the participants will be placed recumbently in a bed. Two cannulas will be inserted in the cubital veins: one for collection of arterialized blood samples and one in the contralateral vein for infusions. The forearm from which blood samples are drawn will be wrapped in a heating blanket (50°C) throughout the experiment. Immediately after taking background samples, a primed constant infusion of [6,6-D2]glucose (D2-glucose) (priming bolus of 40 µmol/kg; continuous infusion rate of 0.4 µmol· min·kg-1) and [1,1,2,3,3,-D5] glycerol (D5-glycerol) (priming bolus of 1.5 µmol/kg; continuous infusion rate 0.1 µmol· min·kg-1) will be started (t=0 min) and maintained for 360 min to determine glucose and glycerol kinetics in the basal and insulin-stimulated state, however the continuous infusion rates will be changed during insulin infusion. The first steady-state period will be defined as the last 30 min of the 120-min basal period, when the tracer equilibria of [D2]glucose and [D5]glycerol are expected; the low grade insulin infusion (10 mU/m2 per min) steady-state period will be defined as the last 30 min of the first insulin clamp period (210-240 min), during which the infusion rate of D2-glucose will be increased to 0.56 µmol· min·kg-1, and the infusion rate of D5-glycerol will be reduced to 0.05 µmol· min·kg-1. The high grade insulin infusion (40 mU/m2 per min) steady-state period will be defined as the last 30 min of the second insulin clamp period (330-360 min), during which the infusion rate of D2-glucose will be increased to 1.0 µmol· min·kg-1, and the infusion rate of D5-glycerol will be reduced to 0.025 µmol· min·kg-1. Following the basal steady-state period at the time point 120 min, a continuous insulin infusion will be initiated and fixed at 10 mU/m2 per min, the infusion rate. At the time point 240 min the continuous insulin infusion will be primed and raised to 40 mU/m2 per min until the time point 360 min. A variable infusion of unlabelled glucose (180 g/l) will be used to maintain euglycemia during insulin infusion. Plasma glucose concentrations will be monitored bedside every 5 min during clamp using the glucose oxidase method (Yellow Springs Instrument Model 2300 STAT plus analyser, Yellow Springs, Ohio, USA). The target plasma glucose concentration will be 5 mM. Blood samples for measuring plasma glucose and glycerol enrichments will be drawn at baseline (0 min) and in the first steady state period (90, 100, 110 and 120 min) and during the insulin-stimulated steady state period (330, 340, 350 and 360 min). All isotopes will be purchased from Cambridge Isotopes Laboratories (Andover, MA). Blood samples for measuring plasma glycerol and lactate will be drawn at baseline and in the first (90 to 120 min), second (210 to 240 min) and third (330-360 min) steady-state period. Samples for determining plasma insulin, C-peptide and glucagon will be drawn at (0, 60, 90, 100, 110, 120, 135, 150, 165, 180, 195, 210, 220, 230, 240, 255, 270, 285, 300, 315, 330, 340, 350, 360 min). Blood samples for determining FFAs, HbA1c, total-, High Density Lipoprotein (HDL)- -, Low Density Lipoprotein (LDL)- and Very Low Density Lipoprotein (VLDL)-cholesterol, and triglycerides will be drawn at baseline, and blood samples for measuring FFAs in the insulin-stimulated state will be drawn at 240 and 360 min. Urine samples will be collected at 0, 120, 240 and 360 min.

Indirect calorimetry will be performed during basal (90-120 min), low (210-240 min) and high grade (330-360 min) insulin-stimulated steady-state to determine oxygen consumption (V02) and carbon dioxide production (VC02). A flow-through canopy gas analyser will be used, as described by (25). The average gas exchange over the three 30-min steady-state periods (basal and insulin-stimulated) will be used to calculate rates of glucose and fat oxidation.

Muscle and fat biopsies will be performed in the end of the basal (t=120 min) and high grade insulin-stimulated (t=360 min) steady-state periods. Muscle and fat biopsies will be obtained under local anaesthesia, from musculi vastus lateralis and subcutaneous abdominal fat using a modified Bergström's needle (including suction) at 120 (basal) and 360 min (high grade insulin-stimulated). Biopsies will be frozen in liquid nitrogen and stored at -80ºC for later analysis. The total amount of extracted tissue will amount to 400-600 mg.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe plaque psoriasis with psoriasis area and severity index (PASI) >8 (exclusively for the patient group)
* Normal fasting plasma glucose (FPG) below 6 mM and haemoglobin A1c (HbA1c) ≤42 mmol/mol(6.0%)
* Normal haemoglobin
* Informed consent

Exclusion Criteria:

* Diabetes (type 1 and type 2 diabetes)
* First degree relatives with diabetes
* Other chronic inflammatory diseases
* Pregnancy or breast feeding
* Psychiatric diseases
* Treatment with drugs that might affect the glucose metabolism within a month prior to the project
* Nephropathy (serum creatinine >130 µM and/or albuminuria)
* Liver disease (alanine aminotransferase (ALT) and/or serum aspartate aminotransferase (AST) >2×normal values)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caucasian adults
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2016-08; Primary Completion 2019-01-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | 6 hours
  Experimental day 2

SECONDARY OUTCOMES:
Non-oxidative glucose metabolism | 6 hours
  Experimental day 2
Endogenous glucose production | 6 hours
  Experimental day 2
Lipolysis | 6 hours
  Experimental day 2
glucose oxidation | 6 hours
  Experimental day 2
Fat oxidation | 6 hours
  Experimental day 2
Molecular changes in muscle and fat tissue | 6 hours
  Experimental day 2
Beta-cell secretion rate | 1 hour
  Experimental day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Denmark, Hellerup, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No